CLINICAL TRIAL: NCT03773380
Title: Breathe Anew: Designing and Testing the Feasibility of a Novel Intervention for Lung Cancer Survivorship
Brief Title: Breathe Anew for Lung Cancer Survivorship
Acronym: BA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: St. Joseph's Healthcare Hamilton (Other)
Responsible Party: Principal Investigator, Wael Hanna, Associate Professor of Surgery, St. Joseph's Healthcare Hamilton
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SJHH-BA
Record Dates: First submitted 2018-12-10; First posted 2018-12-12 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2022-03

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Wearable Electronic Devices

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Feasibility (Experimental): 50 patients will be recruited to take part in this feasibility study. They will all undergo this Breathe Anew Program post-surgery. Breathe Anew consists of radiological surveillance, physical rehabilitation using a Fitbit, mindfulness therapy, and referral for symptom management specialists when needed.
  Interventions: Combination Product: Breathe Anew Survivorship Program

INTERVENTIONS:
Combination Product: Breathe Anew Survivorship Program — The feasibility will be tested of the Breathe Anew Survivorship Program
  Other Names: Wearable Technology, Mindfulness Therapy

SUMMARY:
Survivorship programs have become an integral component of modern cancer care programs. In Canada, there has been tremendous success for survivorship programs for breast, prostate, and colorectal cancer, however lung cancer survivorship programs have not been widely developed. The complexity of the disease, high mortality, short survival times, high cost of surveillance, and patient habits have traditionally been barriers against the success of lung cancer survivorship programs. The investigator proposes a feasibility study to pilot a novel intervention titled Breathe Anew, which will aim to identify and overcome the barriers to the design and implementation of a lung cancer survivorship program. The investigator has assembled a multi-disciplinary team of experts and lung cancer survivors who will develop the Breathe Anew survivorship intervention. The intervention will be vetted using an integrated knowledge translation approach, which will involve members of the target population, primarily patients who previously underwent lung resection, to modify the intervention and ensure acceptability. After Breathe Anew has been designed, it will be tested in a pilot study of 50 patients to ensure its feasibility and determine its cost. The ultimate goal of this feasibility study is to lay the groundwork for a subsequent comparative trial to evaluate the impact of Breathe Anew on patient-important outcomes including health related quality and length of life and postoperative complications.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* All patients at St. Joseph's Healthcare Hamilton who received lung resection for Stage I, Stage II, or Stage IIIa Non-Small Cell Lung Cancer are eligible to enroll.
* Owns a smart device

Exclusion Criteria:

* Patients who received lung resection for Stage IIIb or IV Non-Small Cell Lung Cancer
* Patients with affected mobility (walker, wheelchair)
* Patients who use oxygen at home

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-01-02 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Compliance | 12 months
  The feasibility of Breath Anew, as measured by a rate of compliance of >70% with all the components of the intervention.

SECONDARY OUTCOMES:
Accrual Rate | 12 months
  Rate of accrual to the intervention
Patient-Reported Satisfaction | 12 months
  Using the EQ-5D-5L, which is a standardized instrument developed by the EuroQol Group as a measure of health-related quality of life. The EQ-5D-5L asks the participant to indicate what best describes their health on the day the scale is administered and it consists of 5 dimensions: Mobility, Self-Care, Usual Activities, Pain/Discomfort, and Anxiety/Depression which are measured by a severity scale from 1-5 (no problems = 1, slight problems = 2, moderate problems = 3, severe problems = 4, or completely unable to = 5).
Cost Per Patient | 12 months
  Cost per patient for the duration of the intervention

CONTACTS AND LOCATIONS:
Locations (1):
- St. Joseph's Healthcare Hamilton, Hamilton, Ontario, Canada